CLINICAL TRIAL: NCT04996901
Title: The Chinese ST-Segment Elevation Myocardial Infarction Primary Percutaneous Coronary Intervention Registry
Brief Title: The Chinese STEMI PPCI Registry (CSPR)
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Collaborators: The First College of Clinical Medical Science, China Three Gorges University (Unknown); The First Affiliated Hospital of Dalian Medical University (Other); Jiangxi Provincial People's Hopital (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Xiangyang No.1 People's Hospital (Other); Wuhan Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 958374
Record Dates: First submitted 2021-07-27; First posted 2021-08-09 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- derivation cohort: Data from Renmin Hospital of Wuhan University, The First College of Clinical Medical Science, China Three Gorges University, The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture, Xiangyang No.1 People's Hospital，and Wuhan Third Hospital will be used as a derivation cohort.
  Interventions: Other: no intervention
- validation cohort: Data from The First Affiliated Hospital of Dalian Medical University and Jiangxi Provincial People's Hopital will be used as a derivation cohort.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The purpose of this study is to develop a risk score to predict the risks of in-hospital major adverse cardiac events in ST-segment elevation myocardial infarction patients treated by primary percutaneous coronary intervention.

DETAILED DESCRIPTION:
The CSPR trial is an observational clinical trial to derive and validate a readily useable risk score to identify patients at high risk of in-hospital major adverse cardiac events in 5594 patients presenting with a ST-segment elevation myocardial infarction and treated by primary percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. ST-segment elevation myocardial infarction was defined according to the universal definition of myocardial infarction
3. STEMI treated by pPCI

Exclusion Criteria:

1. Patient with heart failure in admission
2. STEMI with symptom-onset-to-balloon time>24h
3. pPCI was not successful or only underwent coronary angiography
4. Killip class ≥II in admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with STEMI were treated by primary percutaneous coronary intervention at 7 large centers from central China.
Sampling Method: Non-Probability Sample
Enrollment: 5594 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
in-hospital acute de novo heart failure | in-hospital outcome, until discharge
  Killip class ≥II
cardiogenic shock | in-hospital outcome, until discharge
  according to the universal definition
death | in-hospital outcome, until discharge
  according to the universal definition

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Cheng, Study Director — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan university, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Luo D, Lei Y, Hu Z, Tian H, Chen X, Zhou W, Li M, Liu S, Jin X, Wang Y, Zhang B, Zhou Q, Chen J. Correlation between abnormal microvascular perfusion and quantitative flow ratio after primary PCI in patients with STEMI. Int J Cardiol. 2025 Mar 1;422:132949. doi: 10.1016/j.ijcard.2024.132949. Epub 2024 Dec 31. PMID 39746473
- [Derived] Wang H, Yang Y, Zeng P, Huang R, Cai X, Shao L, Liu F, Lei Y, Li D, Fan Z, Yang J, Zhang J, Yang J. Association between Systemic Immune-Inflammation Index (SII) and New-Onset In-Hospital Heart Failure in Patients with STEMI after Primary PCI. Rev Cardiovasc Med. 2024 Oct 24;25(10):382. doi: 10.31083/j.rcm2510382. eCollection 2024 Oct. PMID 39484131
- [Derived] Hu Z, Luo D, Zhou WJ, Xu CW, Chen XZ, Zhang BF, Jin X, Wang Y, Zhang J, Wu H, Liu FY, Lei YH, Li DS, Cai XY, Jiang H, Chen J. Association between admission blood pressure and spontaneous reperfusion and long-term prognosis in STEMI patients: an observational and multicenter study. BMC Cardiovasc Disord. 2024 Sep 18;24(1):500. doi: 10.1186/s12872-024-04168-4. PMID 39294617
- [Derived] Luo D, Huang R, Wang X, Zhang J, Cai X, Liu F, Lei Y, Li D, Zhou W, Xu C, Huang B, Jiang H, Chen J. INTRA-AORTIC BALLOON PUMP REDUCES 30-DAY MORTALITY IN EARLY-STAGE CARDIOGENIC SHOCK COMPLICATING ACUTE MYOCARDIAL INFARCTION ACCORDING TO SCAI CLASSIFICATION. Shock. 2023 Sep 1;60(3):385-391. doi: 10.1097/SHK.0000000000002184. Epub 2023 Aug 4. PMID 37548623